CLINICAL TRIAL: NCT06392607
Title: Euclid Phoenix Lens Design Trial Part 2
Brief Title: Euclid Phoenix Lens Design Trial 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Euclid Systems Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU-PHX-RCT-002
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Myopia; Cornea
MeSH Terms: conditions — Myopia; Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Euclid orthokeartology (standard coating) (Experimental): Euclid Orthokeratology Contact Lenses are lathe cut contact lenses with spherical posterior surfaces. The posterior curve is selected to properly fit an individual eye for orthokeratology and the anterior curve is selected to provide the necessary optical power for a temporary reduction of myopia. A peripheral curve system on the posterior surface allows tear exchange between the lens and the cornea.
  Interventions: Device: Euclid orthokeratology (standard coating)
- Euclid orthokeartology (enhanced coating) (Experimental): Euclid Orthokeratology Contact Lenses are lathe cut contact lenses with spherical posterior surfaces. The posterior curve is selected to properly fit an individual eye for orthokeratology and the anterior curve is selected to provide the necessary optical power for a temporary reduction of myopia. A peripheral curve system on the posterior surface allows tear exchange between the lens and the cornea.
  Interventions: Device: Euclid orthokeratology (enhanced coating)

INTERVENTIONS:
Device: Euclid orthokeratology (standard coating) — Lens with the current coating
  Arms: Euclid orthokeartology (standard coating)
Device: Euclid orthokeratology (enhanced coating) — Lens with the enhanced coating
  Arms: Euclid orthokeartology (enhanced coating)

SUMMARY:
Lens wettability and subjective comfort of Euclid orthokeratology lenses with and without an enhanced coating will be compared in 50 children. Axial elongation will be monitored in pediatric patients who qualify and consent.

DETAILED DESCRIPTION:
The primary objective of this trial is to provide an assessment of the lens wettability and patient comfort with an enhanced surface treatment for the Emerald Lens design when used by practitioners with moderate experience with fitting Euclid orthokeratology lenses.

The hypothesis to be tested is that the proportion of participants with a lens wettability score of > 3 (on a 5 point scale) with the enhanced surface treatment will be greater than that of the current lens surface, using a 1 to 5 scale

The primary outcome variable is lens wettability as measured on eye using a 1 to 5 scale

This clinical investigation will be a prospective, randomized, double-masked two-arm non-crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age or, if under legal age have written consent of their parent or guardian to participate.
* Sign written Informed Consent (and the California Bill of Rights, if applicable).
* Ages 6-35 (inclusive) and able to understand and assent to participation
* Current wearers of Euclid Emerald (Oprifocon A) Orthokeratology lenses, which at initiation of fitting, had

  * Need of optical correction for myopia, from -1.00 to -5.00 Diopters (D).
  * Refractive astigmatism of less than -1.50 D.
* Have a minimum Best Spectacle Corrected Visual Acuity (BSCVA) of 20/40 or better in each eye.
* Have acceptable or optimal fit with study lenses (once fitting has been completed) and be willing to wear these lenses as directed for the duration of the study.
* On examination, have ocular findings considered to be within normal limits, including:

  * No evidence of active infection involving the conjunctiva, lids or adnexa.
  * No evidence of structural abnormalities of the lid, conjunctiva or adnexal tissue considered significant by the investigator to include minimum levels (Grade 2 or less) of tarsal-conjunctival abnormalities
  * Clear corneas with no evidence of edema, staining, opacities, corneal neovascularization greater than a trace amount (i.e. All vessels extending less than 1.5 mm from the limbus); all as observed on slit lamp examination.
  * No iritis.
  * No herpes keratitis (recurrent or otherwise) or other active ocular disease that would contraindicate lens wear or lessen attainability of VA sought in this study (20/40 or better).
  * No evidence of dry eye or meibomian gland dysfunction
* Normal binocularity (no amblyopia or strabismus, and no anisometropia of greater than 2.00D)
* Be willing and able to follow instructions and attend the schedule of follow-up visits.

Exclusion Criteria:

* Does not meet the any of the above inclusion criteria
* Not able or willing to provide informed consent and assent
* Requires concurrent ocular medication
* Eye injury or surgery within twelve weeks immediately prior to enrollment
* Pre-existing ocular condition that would preclude contact lens fitting
* Currently enrolled in an ophthalmic clinical trial
* Pregnant or lactating or expect to become pregnant during the trial
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Allergy or sensitivity to any product used in this trial
* Any systemic disease including autoimmune disease, immunocompromising diseases, connective tissue disease, clinically significant atopic diseases, insulin dependent diabetes, use of medications including corticosteroids and antimetabolites that may affect the eye or be exaggerated by contact lenses.
* Strabismus/amblyopia
* Habitual uncorrected anisometropia ≥ 2.00D
* Subjects who have undergone corneal refractive surgery
* Subjects with severe corneal irregularity contraindicating lens wear
* Inability to wear contact lenses, or an unacceptable contact lens fit
* Poor or unacceptable fit with any study lens
* Employees, staff or family members of personnel at the site

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Lens wettability | 12 months
  Lens wettability as measured on eye using a 1 to 5 scale

SECONDARY OUTCOMES:
Patient comfort ratings | 12 months
  Patient comfort as measured by patient reported outcome using a 1 to 5 scale

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Pinecone Vision Center, Sartell, Minnesota
  - Somerset Eye Care, North Brunswick, New Jersey
  - Southern College of Optometry, Memphis, Tennessee
  - Specialty Eyecare Group, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: Undecided